CLINICAL TRIAL: NCT06841211
Title: Optimizing Prostate Biopsy Schemes in Men With Multiple mpMRI Visible Lesions: a Randomized Controlled Trial Evaluating the Efficacy of Perilesional/Regional Biopsy in Prostate Cancer Diagnosis Among Men With Multiple mpMRI Visible Lesions
Brief Title: Optimizing Prostate Biopsy Schemes in Men With Multiple mpMRI Visible Lesions
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Responsible Party: Principal Investigator, LIU Yi, Associate chief physician, Peking University First Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: PB-03
Record Dates: First submitted 2025-02-18; First posted 2025-02-24 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; Randomized controlled trial; Targeted biopsy; Perilesional biopsy; Diagnosis
MeSH Terms: conditions — Prostatic Neoplasms; Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Targeted and perilesional biopsy (TPLBx) (Experimental): For patients in the TPLBx group, two-core targeted biopsies (TBs) were obtained within each predefined mpMRI suspicious lesion (region of interest, ROI), followed by ring-distributed four cores within a 10-15 mm radius around the ROI. The location of these cores depended on the shape and location of the ROI.
  Interventions: Procedure: Targeted and perilesional biopsy (TPLBx)
- Combined targeted and systematic biopsy (CTSBx) (Experimental): For patients in the CTSBx group, two-core TBs from the lesion were performed within each ROI, followed by a sextant 12-core systematic biopsy (SB).
  Interventions: Procedure: Combined targeted and systematic biopsy (CTSBx)

INTERVENTIONS:
Procedure: Targeted and perilesional biopsy (TPLBx) — The biopsy procedure is conducted by highly skilled and experienced urologists who specialize in performing prostate biopsies. A single dose of prophylactic antibiotics (usually cephalosporins) is routinely administered following a test dose 30 min before the procedure. Each patient is placed in the lithotomy position. Povidone-iodine is routinely used to clean perineum before the biopsy. The MRI-TRUS biopsy system is iFUSS (image fusion surgical system, Carbon Med), consisting of a 3D reconstruction and planning software (Carbon Med) and a bi-planar TRUS probe (ECL8-4-B, Carbon Med). Color Doppler examination is performed from the base to the apex. For each predefined mpMRI suspicious lesion, two-core TBs are obtained within the ROI, followed by ring-distributed four cores within a 10-15 mm radius around the ROI. The location of these cores depends on the shape and location of the suspicious lesion.
  Arms: Targeted and perilesional biopsy (TPLBx)
Procedure: Combined targeted and systematic biopsy (CTSBx) — The biopsy procedure is conducted by highly skilled and experienced urologists who specialize in performing prostate biopsies. A single dose of prophylactic antibiotics (usually cephalosporins) is routinely administered following a test dose 30 min before the procedure. Each patient is placed in the lithotomy position. Povidone-iodine is routinely used to clean perineum before the biopsy. The MRI-TRUS biopsy system is iFUSS (image fusion surgical system, Carbon Med), consisting of a 3D reconstruction and planning software (Carbon Med) and a bi-planar TRUS probe (ECL8-4-B, Carbon Med). Color Doppler examination is performed from the base to the apex. Two-core TBs from the lesion were performed within each predefined mpMRI suspicious lesion, followed by fore-zone 12-core biopsy.
  Arms: Combined targeted and systematic biopsy (CTSBx)

SUMMARY:
The goal of this randomized controlled trial (RCT) is to evaluate the efficacy of different prostate biopsy schemes in prostate cancer diagnosis among men with multiple mpMRI visible lesions, including combination of targeted and perilesional/regional biopsy (PB/RB) (TPLBx) and combination of systematic biopsy and targeted biopsy (CTSBx).

The main questions it aims to answer are:

Does TPLBx promote the accurate diagnosis of clinically significant prostate cancer (csPCa) among men with multiple mpMRI visible lesions? What's the value of TPLBx in improving the evaluation of prostate cancer when developing the treatment plan for patients with multiple mpMRI visible lesions? What's the value of TPLBx in avoiding the adverse pathological outcomes after the radical prostatectomy such as upgrade, upstage, capsule invasion, and positive surgical margin among patients with multiple mpMRI visible lesions? Researchers will compare the cancer detection rates of TPLBx and CTSBx to explore the efficacy of different prostate biopsy schemes. They will evaluate the occurrence rates of adverse pathological changes of different prostate biopsy schemes after the radical prostatectomy (RP).

Participants will:

Receive TPLBx or CTSBx.

DETAILED DESCRIPTION:
Prostate biopsies have been the cornerstone of prostate cancer (PCa) diagnosis, risk stratification, and treatment planning. The optimal biopsy scheme should achieve the highest csPCa detection rates with the most accurate core sites and the least biopsy-cores. The combined targeted and systematic biopsy (CTSBx) could effectively detect clinically significant PCa (csPCa) and was the standard scheme for patients with visible suspicious lesions on multiparametric MRI (mpMRI) in the past. However, some limitations existed in the CTSBx scheme, including the detection of clinically insignificant PCa (ciPCa), the risk of post-biopsy complications, and adverse pathological changes such as upgrade, upstage, capsule invasion, and positive surgical margin after the radical prostatectomy (RP). Therefore, more and more radiologists and urologists focused on the issue of optimization of prostate biopsy schemes. Recent studies demonstrated that the majority of csPCa were found within a band of 10-mm radius outside MRI lesions (the penumbra). Focusing biopsy cores within and around the region of interest (ROI), known as targeted and perilesional biopsy (TPLBx) scheme, is recommended by the latest EAU guideline for the diagnosis of patients with visible suspicious lesions on multiparametric MRI (mpMRI).

Prostate cancer generally occurs multifocally. The incidence of multiple lesions among different cohorts in previous studies ranges between 20% and 50%. Though the CTSBx schemes are usually utilized for these patients, some previous studies suggested that additional systematic biopsy is of limited informative value in terms of overall csPCa detection. Therefore, the optimal prostate biopsy scheme for patients with multiple visible mpMRI suspicious lesions is still a matter of debate. Compared with the CTSBx scheme, the TPLBx changed the distribution of the biopsy-core according to the location of visible suspicious lesions. Many studies have preliminarily verified that the diagnostic efficacy of TPLBx was not inferior to that of CTSBx with the benefits of decreasing the detection of ciPCa and reducing biopsy cores. TPLBx scheme focuses biopsy cores within and around the ROI, which may evaluate the pathological characteristics of mpMRI visible suspicious lesions more accurately, benefiting for the treatment planning and reducing the occurrence rates of adverse pathological changes after the radical prostatectomy (RP). However, current data for TPLBx schemes are mostly retrospective, and few studies focused on the application of TPLBx for patients with multiple mpMRI visible lesions. Thus, this randomized controlled trial (RCT) aims to evaluate the efficacy of TPLBx and CTSBx schemes for patients with multiple mpMRI visible lesions, provide high-quality evidence for the optimization of prostate biopsy schemes.

The main questions it aims to answer are:

Does TPLBx promote the accurate diagnosis of clinically significant prostate cancer (csPCa) among men with multiple mpMRI visible lesions? What's the value of TPLBx in improving the evaluation of prostate cancer when developing the treatment plan for patients with multiple mpMRI visible lesions? What's the value of TPLBx in avoiding the adverse pathological outcomes after the radical prostatectomy such as upgrade, upstage, capsule invasion, and positive surgical margin among patients with multiple mpMRI visible lesions? Researchers will compare the cancer detection rates of TPLBx and CTSBx to explore the efficacy of different prostate biopsy schemes. They will evaluate the occurrence rates of adverse pathological changes of different prostate biopsy schemes after the radical prostatectomy (RP).

Participants will:

Receive TPLBx or CTSBx.

ELIGIBILITY:
Inclusion Criteria:

* the age of the patient is between 18 and 85;
* no previous biopsy;
* presence of multiple multiparametric magnetic resonance imaging (mpMRI) visible lesions;
* every mpMRI visible lesion is in accordance with the EAU guidelines for performing perilesional biopsy (PB) (PI-RADS ≥4 or PI-RADS =3, clinical suspicion of PCa);
* a verified prostate-specific antigen (PSA) less than 50 ng/ml;
* complete mpMRI data, and high mpMRI quality (Prostate Imaging Quality [PI-QUAL] V1.0 score ≥3);
* the time interval between prostate biopsy and prostate mpMRI examination should not exceed one month;
* patients with complete prostate biopsy pathological results;
* patients with complete clinical information.

Exclusion Criteria:

* contraindication for mpMRI examination (i.e., in acute attack period such as high fever, coma, epilepsy, prone to cardiac arrest, claustrophobia, presence of ferrous metallic implants, or claustrophobia);
* contraindication for prostate biopsy ((a) in the period of acute infection or fever; (b) hypertensive crisis; (c) in the decompensated stage of heart failure; (d) diseases with severe bleeding tendency; (e) poorly controlled complications of hypertension or diabetes; (f) patients with severe internal or external hemorrhoids, perianal or rectal lesions should not undergo transrectal biopsy);
* a history of radiotherapy, chemotherapy, androgen deprivation therapy, or surgery for PCa;
* patients with previous biopsy;
* the absence of MRI-visible prostate lesions or presence of single suspicious lesions;
* PI-RADS V2.1 <3;
* unqualified or incomplete mpMRI data;
* the patient could not cooperate to complete the prostate biopsy;
* the patients or their family members refused to participate in this study;
* patients with incomplete clinical information.

Ages: 18 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-02-01 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
The clinically significant prostate cancer (csPCa) detection rate for TPLBx and CTSBx schemes | One month after the biopsy procedure.
  The csPCa was defined as prostate cancer (PCa) with a grade group ≥2 or Gleason score (GS) ≥3+4. The reference standard was the pathological result.

SECONDARY OUTCOMES:
The PCa detection rate | One month after the biopsy procedure.
  The PCa detection rate for TPLBx and CTSBx schemes.
The clinically insignificant PCa (ciPCa) detection rate | One month after the biopsy procedure.
  The ciPCa was defined as PCa with a grade group <2 or GS <3+4. The reference standard was the pathological result.
The higher-grade PCa detection rate for TPLBx and CTSBx schemes | One month after the biopsy procedure.
  The higher-grade PCa was defined as PCa with a grade group ≥3 or GS≥4+3. The reference standard was the pathological result.
The Gleason score (GS) of the biopsy sample | One month after the biopsy procedure.
  The Gleason score was reported by senior uropathologists according to the Standards of Reporting for MRI Targeted Biopsy Studies (START) criteria and interpreted according to the recommendations of the International Society of Urological Pathology (ISUP) Grade Group.
The GS of radical prostatectomy (RP) specimens | One month after the RP.
  The overall grade was assigned based on the part with the highest Gleason score according to the recommendations of the ISUP. For the RP specimens, the overall grade was assigned based on the part with the highest Gleason score according to the recommendations of the ISUP.
The adverse pathological outcomes of radical prostatectomy (RP) specimens | One month after the RP.
  The adverse pathological outcomes such as upgrading, upstaging, positive surgical margin, and capsule invasion were assessed and reported by the senior uropathologists based on RP specimens.

CONTACTS AND LOCATIONS:
Overall Officials: Yi LIU, Principal Investigator — Peking University First Hospital
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No